CLINICAL TRIAL: NCT06409234
Title: EuPreCHO: European Study on Perioperative Management and Outcome Following Preoperative Transthoracic Echocardiography in Noncardiac Surgery Patients
Brief Title: Perioperative Management & Outcome Following Preoperative Transthoracic Echocardiography in Noncardiac Surgery Patients
Status: Not yet recruiting | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: EuPreCHO
Record Dates: First submitted 2024-04-08; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-04

CONDITIONS: Elective Surgical Procedure
Keywords: transthoracic echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exposed group: 5500 exposed group will be patients in whom Transthoracic Echocardiography was performed within 3 months before surgery. Controls will be patients in whom Transthoracic Echocardiography was NOT performed.
  Interventions: Other: Transthoracic Echocardiography Recieved

INTERVENTIONS:
Other: Transthoracic Echocardiography Recieved — Transthoracic Echocardiography Recieved

SUMMARY:
In August 2022 the European Society of Cardiology published updated guidelines including recommendations on preoperative transthoracic echocardiography. The update resulted in broadened criteria for preoperative transthoracic echocardiography. The impact of preoperative transthoracic echocardiography on outcome is controversial and the evidence was mostly derived from administrative databases. Also there is also a knowledge gap in terms of what changes in perioperative managements are derived from transthoracic echocardiography information in current daily practice in Europe and what their impact on outcome may be. Further, a secondary analysis in a large international cohort suggests that the criteria endorsed by the guidelines to define the class of recommendation of transthoracic echocardiography may not be efficient.

DETAILED DESCRIPTION:
The target population consists of patients at elevated cardiovascular risk undergoing elective, intermediate or high-risk noncardiac surgery. The planned sample size is 5500 exposed and 2750 non-exposed

ELIGIBILITY:
Inclusion Criteria

* aged ≥65 years OR
* above 18 years and presenting ≥2 cardiovascular risk factors (hypertension, smoking, dyslipidaemia, diabetes, family history of CVD) OR
* above 18 years with known cardiovascular disease

Exclusion Criteria

* under 18 years of age
* day surgery
* urgent/emergency procedures
* current ICU patient (i.e. in ICU on day-1 or the day of the index surgery (day 0)),
* cardiac surgery within the last month prior according to the index noncardiac procedure (of note this does not include cardiological interventions like TAVI or valvuloplasty),
* unwilling or unable to provide informed consent,
* unable to complete the WHODAS questionnaire (literacy or language barrier)
* Previous enrollment in EuPreCHO (in case of repeated surgery)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: EuPreCHO is a prospective, international, case control study. RQ3 will be assessed in a cohort consisting of the cases only. Any hospital in Europe (as defined by the World Health Organisation) is welcome to participate as a study centre. Study centre registration occurs online via the dedicated Call for Centres form on the ESAIC website. Centres will be asked to enroll a minimum of 50 cases and 25 controls within the 12-month period planned for EuPreCHO enrollment. Within the enrollment period, the start of recruitment for individual centres is at the discretion of the local PI, provided that there is a prior IRB approval. Recruitment across all centres will continue until enrollment of the planned sample size.
Sampling Method: Non-Probability Sample
Enrollment: 8250 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathology | 30 days
  Decreased contractility (LVEF ≤40% by Simpson's method or eyeballing) or based on corresponding qualitative statement in TTE report. Significant LV diastoic: E/A <0.8 + E>50cm/sec OR E/A >0.8 to <2 + at least ≥ 2 additional criteria ( Average E/e' ratio >14, peak TR velocity >2,8 m/sec, LA volume index >34 mL/m2.

SECONDARY OUTCOMES:
Disability-free survival at 30 days | 30 days
  WHODAS scale-none=0 to extreme=4, for a total maximal score of 48 and transformed into the percentage of maximal disability score

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Lurati Buse, Prof, Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (1):
- University Hospital Düsseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No